CLINICAL TRIAL: NCT04000282
Title: An Open-label, First-in-human, Single Agent, Dose-escalation and Expansion Study for the Evaluation of Safety, Pharmacokinetics, Pharmacodynamics and Anti-tumor Activity of SAR442085 in Patients With Relapsed or Refractory Multiple Myeloma (RRMM)
Brief Title: First-in-human Single Agent Study of SAR442085 in Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TED16132; U1111-1223-4410 (Registry Identifier: ICTRP); 2019-001018-40 (EudraCT Number)
Record Dates: First submitted 2019-06-11; First posted 2019-06-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: SAR442085 dose escalation (Experimental): SAR442085 will be given intravenously weekly for 4 weeks (Cycle 1) and on Day 1 and Day 15 of each subsequent cycle until the patient has progressive disease, unacceptable toxicity or other reasons to terminate study treatment. Each cycle will be approximately 28 days in duration.
  Interventions: Drug: SAR442085
- Part B: SAR442085 dose expansion (Experimental): SAR442085 will be given intravenously weekly for 4 weeks (Cycle 1) and on Day 1 and Day 15 of each subsequent cycle until the patient has progressive disease, unacceptable toxicity or other reasons to terminate study treatment. Each cycle will be approximately 28 days in duration.
  Interventions: Drug: SAR442085

INTERVENTIONS:
Drug: SAR442085 — Pharmaceutical form:Sterile lyophilized powder for reconstitution for infusion Route of administration: intravenous

SUMMARY:
Primary Objectives:

* Dose Escalation Part A: To determine the maximum tolerated dose (MTD) of SAR442085 administered as a single agent in patients with relapsed or refractory multiple myeloma (RRMM), and determine the recommended Phase 2 dose (RP2D) for the subsequent Expansion Part B
* Dose Expansion Part B: To assess the antitumor activity of single agent of SAR442085 at the RP2D in patients with RRMM

Secondary Objectives:

* To characterize the safety profile of SAR442085
* To characterize the pharmacokinetics (PK) profile of SAR442085 when administered as a single agent
* To evaluate the potential immunogenicity of SAR442085
* To assess preliminary evidence of antitumor activity in the Dose Escalation Part A

DETAILED DESCRIPTION:
Patient will continue to receive study medication until disease progression, unacceptable toxicity, withdrawal of informed consent, or other reason why investigator considers it appropriate to discontinue study medication. Once permanently discontinued, study medication cannot be restarted at later timepoint.

ELIGIBILITY:
Inclusion criteria :

* Participant must be at least 18 years of age or of the country's legal age of majority if the legal age is >18 years old, at the time of signing the informed consent.
* Participant has given voluntary written informed consent.
* Participant has been previousy diagnosed with multiple myeloma based on standard criteria.
* Part A: (1) participant has received at least 3 prior lines of therapy for multiple myeloma, or at least 2 prior lines of therapy if at least 1 of those lines consisted of 2 or more multi-agent regimens (eg, multi-agent induction regimen with autologous stem cell transplantation, followed by maintenance regimen). (2) Prior therapy for multiple myeloma has included at least 1 proteasome inhibitor (bortezomib, carfilzomib, ixazomib), at least 1 immunomodulatory agent (lenalidomide, thalidomide, pomalidomide), at least 1 anti-CD38 monoclonal antibody and at least 1 steroid. Applicable countries in EU and Asia can enroll anti-CD38 naive RRMM patients from DL4 and onwards. (3) Participant had at least a minimal response (MR) to the anti-CD38 antibody containing regimen and had last dose of anti-CD38 monoclonal antibody at least 9 months prior to study entry. Applicable countries in EU and Asia can enroll anti-CD38 naive RRMM patients from DL4 and onwards.
* Part B and the last cohort(s) of Part A: (1) participant has received at least 3 prior lines of therapy for multiple myeloma, or at least 2 prior line of therapy if at least 1 of those lines consisted of 2 or more multi-agent regimens (eg, multi-agent induction regimen with autologous stem cell transplantation, followed by maintenance regimen). (2) Prior therapy for multiple myeloma has included at least 1 proteasome inhibitor (bortezomib, carfilzomib, ixazomib), at least 1 immunomodulatory agent (lenalidomide, thalidomide, pomalidomide) and at least 1 steroid. (3) Prior therapy has not included an anti-CD38 monoclonal antibody.
* Participant has myeloma disease progression on or after last therapy.
* Participant must have measurable disease as defined as at least one of the following:

  * Serum M protein ≥0.5 g/dL (≥5 g/L)
  * Urine M protein ≥200 mg/24 hours
  * Serum FLC assay: Involved FLC assay ≥10 mg/dL (≥100 mg/L) and an abnormal serum
  * FLC ratio (<0.26 or >1.65).
* A male participant must agree to use contraception during the intervention period and for at least 150 days after the last dose of study drug and refrain from donating sperm during this period.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP)
  * A WOCBP who agrees to follow the contraceptive guidance during the intervention period and for at least 150 days after the last dose of study intervention.

Exclusion criteria:

* Participant is diagnosed or treated for another malignancy within 3 years prior to enrollment, with the exception of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, superficial bladder carcinoma or low risk prostate cancer.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status score >2.
* Participant has a history of Chronic obstructive pulmonary disease (COPD) or asthma.
* Participant has not recovered from adverse reactions to prior myeloma treatment or procedures (chemotherapy, immunotherapy, radiation therapy) to NCI CTCAE Grade ≤1 or baseline (exception: alopecia).
* Participant has congestive heart failure (New York Heart Association) Grade ≥II; cardiac myopathy, active ischemia, or any other uncontrolled cardiac condition such as angina pectoris, clinically significant arrhythmia requiring therapy including anticoagulants, or clinically significant uncontrolled hypertension, QT interval corrected by the Fridericia method >480 msec (Grade ≥2).
* Participant has had acute myocardial infarction within 6 months before first dose of study medication.
* Participant has ongoing sensory or motor neuropathy of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade ≥3.
* Participant has active autoimmune disease including autoimmune hemolytic anemia, idiopathic thrombocytopenic purpura, inflammatory bowel syndrome, pneumonitis or any chronic condition requiring a higher corticosteroid systemic equivalent than prednisone 10 mg daily.
* Known acquired immunodeficiency syndrome (AIDS) or related illnesses or human immunodeficiency virus (HIV) disease requiring antiretroviral treatment, or to have active hepatitis A, B (defined as a known positive hepatitis B surface antigen (HBsAg) result or positive HepB DNA), or C (defined as a known quantitative hepatitis C [HCV] ribonucleic acid RNA results greater than the lower limits of detection of the assay or positive HCV antigen) infection.
* Participant has positive Coombs test at baseline.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) of SAR442085 (Part A) | At the end of Cycle 1 (each cycle is approximately 28 days)
  MTD is defined as the dose level with highest probability of investigational medicinal product (IMP) related dose limiting toxicity (DLT) rate within the target range (16 to 33%) among dose levels with less than 0.25 probability of DLT rate above target (>33%)
Recommended Phase 2 dose (RP2D) (Part A) | At the end of Cycle 1 (each cycle is approximately 28 days)
  RP2D is defined as the dose selected for the further single agent testing - including in Phase 1 expansion part B.
Overall response rate (Part B) | approximately 6 months after the last patient has started treatment in Part B (approx. 2 years)
  Overall response rate (ORR): is defined as the proportion of patients with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR), using the International Myeloma Working Group (IMWG) criteria.

SECONDARY OUTCOMES:
Treatment-emergent adverse events (AEs)/serious adverse events (SAE) (Both Part A and B) | From baseline to end of treatment + 30 days (approx. 2 years)
  Number of participants with Treatment-Emergent Adverse events (TEAEs) from baseline to End of Study.
PK parameters of SAR442085: Cmax (Both Part A and B) | Cycle 1 Day 1 to Day 28
  Maximum plasma concentration observed (Cmax).
PK parameters of SAR442085: Tmax (Both Part A and B) | Cycle 1 Day 1 to Day 28
  First time to reach Cmax (tmax).
PK parameters of SAR442085: AUC (Both Part A and B) | Cycle 1 Day 1 to Day 28
  Area under the plasma concentration versus time curve extrapolated to infinity (AUC).
Anti-drug antibody (ADA) against SAR442085 (Both Part A and B) | Cycle 1, 2, 3, 6 and 9 (each cycle is approximately 28 days)
  Number of participants with ADA against SAR442085.
Progression-free survival (Part B) | approximately 12 months after the last patient has started treatment in Part B (approx. 2 years)
  Progression-free survival (PFS) is defined as the time interval from the date of enrollment to the date of documented tumor progression as per IMWG or death (due to any cause), whichever comes first.
Duration of response (Part B) | approximately 12 months after the last patient has started treatment in Part B (approx. 2 years)
  Duration of response (DOR) is defined as the time from first documented evidence of CR or PR until progressive disease (PD) as per IMWG or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (12):
- United States (5):
  - City of Hope Site Number : 8400002, Duarte, California
  - Dana Farber Cancer Institute Site Number : 8400003, Boston, Massachusetts
  - Mayo Clinic of Rochester Site Number : 8400005, Rochester, Minnesota
  - UNC Chapel Hill Site Number : 8400006, Chapel Hill, North Carolina
  - Froedtert Hospital & Medical College of Wisconsin Site Number : 8400004, Milwaukee, Wisconsin
- Czechia (3):
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2030003, Ostrava - Poruba
  - Investigational Site Number : 2030001, Prague
- Investigational Site Number : 2500001, Toulouse, France
- Investigational Site Number : 3000001, Athens, Greece
- Investigational Site Number : 7240001, Salamanca, Salamanca, Spain
- Investigational Site Number : 1580001, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Kapoor P, Nathwani N, Jelinek T, Pour L, Perrot A, Dimopoulos MA, Huang SY, Spicka I, Chhabra S, Lichtman E, Mateos MV, Kanagavel D, Zhao L, Guillemin-Paveau H, Mace S, van de Velde H, Richardson PG. An open-label, first-in-human, single agent, dose escalation study for the evaluation of safety and efficacy of SAR442085 in patients with relapsed or refractory multiple myeloma. Eur J Haematol. 2024 Nov;113(5):593-605. doi: 10.1111/ejh.14270. Epub 2024 Jul 12. PMID 38993150
- See also: TED16132 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25358&tenant=MT_SNY_9011